CLINICAL TRIAL: NCT02503137
Title: A Phase 2, Multicenter, Randomized, Double-Blind Study of SM04554 Applied Topically to the Scalp of Male Subjects With Androgenetic Alopecia (AGA) Analyzed by Biopsy of the Scalp Prior To and Post Dosing
Brief Title: A Study of SM04554 Applied Topically to the Scalp of Male Subjects With Androgenetic Alopecia Analyzed by Biopsy of the Scalp Prior To and Post Dosing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04554-AGA-04
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Androgenetic Alopecia
Keywords: male pattern baldness; SM04554; AGA
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental Arm 1 (Experimental): Topical SM04554 0.15% solution, once daily for approximately 90 days
  Interventions: Drug: Topical SM04554 solution
- Experimental Arm 2 (Experimental): Topical SM04554 0.25% solution, once daily for approximately 90 days
  Interventions: Drug: Topical SM04554 solution
- Vehicle (Placebo Comparator): Topical vehicle solution, once daily for approximately 90 days
  Interventions: Drug: Topical Vehicle solution

INTERVENTIONS:
Drug: Topical SM04554 solution
  Arms: Experimental Arm 1; Experimental Arm 2
Drug: Topical Vehicle solution
  Arms: Vehicle

SUMMARY:
This study will assess the safety, tolerability, and efficacy of SM04554 at concentrations of 0.15% and 0.25%. Improved knowledge of the changes in hair counts and immunohistochemical analysis associated with androgenetic alopecia (AGA) before and after treatment with SM04554 and compared to placebo may lead to a greater understanding of the underlying mechanisms of action of SM04554.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AGA with Norwood-Hamilton Classification score of 4, 5, 5A, 5V, or 6
* In good general health, as determined by the Investigator
* Willing and able to attend all study visits
* Willing to undergo two punch biopsies of the scalp
* Willing to inform females, with whom they may interact, that they are using a topical investigational product and direct contact should be avoided as potential harm to a fetus is unknown
* Willing to not use permanent or semi-permanent hair products (e.g., color, texturizers, relaxers) for the duration of the study; daily styling products will be allowed on non-study visit days (e.g., hair gel, mousse, styling spray)
* Willing to use sponsor-supplied shampoo and conditioner in place of regular shampoo and conditioner, for the duration of the study; use of sponsor-supplied conditioner is optional for subjects who do not use conditioner

Exclusion Criteria:

* Clinical diagnosis of alopecia areata or other non-AGA forms of alopecia
* Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
* Males who are sexually active and have a partner who is capable of becoming pregnant, neither of whom have had surgery to become sterilized, that are not using a highly effective method of birth control and are not willing to use a highly effective method of birth control during the study treatment period until 90 days post last dose of study medication
* Current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, seborrheic dermatitis, actinic keratosis), cuts and/or abrasions on the scalp or hands or condition (e.g., sunburn, tattoos) on the treatment area or hands that, in the opinion of the Investigator, might put the subject at risk or interfere with the study conduct or evaluations
* History of or current skin cancer (e.g., melanoma, basal cell carcinoma, squamous cell carcinoma) located anywhere on the body
* History of surgical correction of hair loss on the scalp
* Previous exposure to SM04554
* Use of blood thinners (e.g., Coumadin, Plavix, Lovenox, and aspirin >81mg); low dose aspirin (e.g., ≤81 mg) is allowable
* Use of any products or devices clinically proven to promote scalp hair growth (e.g., finasteride or minoxidil) within 24 weeks prior to study start
* Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, cimetidine) within 12 weeks prior to study start
* Use of semi-permanent hair products (e.g., color, texturizers, relaxers) within 30 days prior to study start
* Use of medicated shampoo or conditioner (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the-counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth) within 30 days prior to study start
* History of hair transplants
* Current use of an occlusive wig, hair extensions, or hair weaves
* Participation in any other investigational drug or medical device trial which included administration of an investigational study medication or medical device, within 30 days or 5 half-lives of the investigational agent, whichever is longer, prior to study start
* Poor peripheral venous access
* Subjects unwilling to refrain from sperm donation during the study treatment period until 90 days post last dose of study medication
* Subjects with pregnant partners at study start
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or are directly affiliated with the study at the investigative site
* Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in number of terminal hair follicles | Baseline and Day 91
  Scalp biopsies obtained prior to initiating therapy and after 90 days of therapy will be compared to determine the change in number of terminal hair follicles over the treatment period.
Change in number of anagen hair follicles | Baseline and Day 91
  Scalp biopsies obtained prior to initiating therapy and after 90 days of therapy will be compared to determine the change in number of anagen hair follicles over the treatment period.
Change in number of telogen hair follicles | Baseline and Day 91
  Scalp biopsies obtained prior to initiating therapy and after 90 days of therapy will be compared to determine the change in number of telogen hair follicles over the treatment period.
Change in number of catagen hair follicles | Baseline and Day 91
  Scalp biopsies obtained prior to initiating therapy and after 90 days of therapy will be compared to determine the change in number of catagen hair follicles over the treatment period.
Change in number of vellus (vellus-like) miniaturized hair follicles | Baseline and Day 91
  Scalp biopsies obtained prior to initiating therapy and after 90 days of therapy will be compared to determine the change in number of vellus (vellus-like) miniaturized hair follicles over the treatment period.
Change in number of indeterminate hair follicles | Baseline and Day 91
  Scalp biopsies obtained prior to initiating therapy and after 90 days of therapy will be compared to determine the change in number of indeterminate hair follicles over the treatment period.

SECONDARY OUTCOMES:
Change in number of terminal hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in the number of terminal hair follicles over the treatment and off-treatment periods.
Change in number of anagen hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in the number of anagen hair follicles over the treatment and off-treatment periods.
Change in number of telogen hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in the number of telogen hair follicles over the treatment and off-treatment periods.
Change in number of catagen hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in the number of catagen hair follicles over the treatment and off-treatment periods.
Change in number of vellus (vellus-like) miniaturized hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in the number of vellus (vellus-like) miniaturized hair follicles over the treatment and off-treatment periods.
Change in number of indeterminate hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in the number of indeterminate hair follicles over the treatment and off-treatment periods.
Change in density of hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in density of hair follicles over the treatment and off-treatment periods.
Ratio of terminal to miniaturized hair follicles (indeterminate hair and vellus hair follicles) | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be used to determine the ratio of terminal to miniaturized hair follicles during the treatment and off-treatment periods.
Change in nuclear expression of beta-catenin | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in nuclear expression of beta-catenin over the treatment and off-treatment periods.
Change in Ki-67 index in epidermis and hair follicles | Baseline, Day 91 and Day 135
  Scalp biopsies obtained prior to initiating therapy, after 90 days of therapy, and after an additional 45 days off therapy will be compared to determine the change in Ki-67 index in epidermis and hair follicles over the treatment and off-treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (5):
- United States (5):
  - Research Site, Clinton Township, Michigan
  - Research Site, Cleveland, Ohio
  - Research Site, College Station, Texas
  - Research Site, Houston, Texas
  - Research Site, Lynchburg, Virginia